CLINICAL TRIAL: NCT05905419
Title: Neurobiological Consequences of Long-Term Opioid Therapy in the Brain and Spinal Cord
Brief Title: Neuroimaging of Opioid Phase (OPAL)
Acronym: OPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00110253; 1R01DA055850 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Opioid Use
Keywords: fibromyalgia; women; brain; functional MRI; opioid; opiate; narcotic; chronic pain; pain
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Female adults with chronic pain who take prescribed opioid medications (Experimental): Opioid taking participants will undergo two study visits, one for each opioid phase ("peak" or "trough")
  Interventions: Other: Opioid Phase
- Female adults with chronic pain who do not take opioid medications (No Intervention): Participants with chronic pain who are not taking opioids will undergo one study visit
- Healthy controls (No Intervention): Healthy female participants who are not taking opioids will undergo one study visit

INTERVENTIONS:
Other: Opioid Phase — Opioid-taking patients are assigned to take their prescribed opioid medication before ("peak" opioid phase) during 1 scan and after ("trough" opioid phase) during the other MRI scan
  Arms: Female adults with chronic pain who take prescribed opioid medications

SUMMARY:
The purpose of this study is to compare activity in the brains of female adults with chronic pain and/or opioid use, and healthy female adults that may help to develop new and targeted treatments for adults with chronic pain and alternatives to opioid therapy.

DETAILED DESCRIPTION:
The objective of the study is to determine differences in neurophysiology and behavior during different phases of opioid use in patients. Study activities will include neuroimaging (MRI and fMRI), behavioral tasks, sensory testing, blood draws, and questionnaires. The neuroimaging data will be analyzed using specialized software; data from questionnaires, sensory testing, and behavioral task performance will be analyzed using standard statistical software. Risks and safety concerns include standard, minimal risks associated with MRI scans, sensory testing, blood draws, and confidentiality.

ELIGIBILITY:
Inclusion Criteria for Healthy Controls:

1. female and ages 18+
2. ability to read/understand English and give consent to participate
3. no current or history of chronic pain
4. not regularly taking any pain-relieving or mood-altering medications (per PI discretion)
5. absence of use of opioid medications

Inclusion Criteria for Individuals with Chronic Pain:

1. female and ages 18 +
2. ability to read/understand English and give consent to participate
3. self-reported or physician diagnosis of fibromyalgia and/or chronic pain
4. current use of opioid medication(s) for inclusion in the opioid patient group -OR- absence of use of opioid medications for inclusion in the non-opioid patient group

Exclusion Criteria (for both groups):

1. limited ability to participate fully in behavioral tasks, longitudinal follow-up
2. MRI contraindication
3. any factors that at the discretion of the investigators would adversely affect the participant or the integrity of the study
4. male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Characterize brain fMRI-based activity related to neurobiological consequences of opioid therapy | During study visits up to 4 weeks apart
  Compare brain fMRI-based response to reward stimuli during a monetary incentive delay (MID) task and functional connectivity of brain reward circuitry during resting state.

SECONDARY OUTCOMES:
Characterize spinal cord fMRI-based activity related to neurobiological consequences of opioid therapy | During study visits up to 4 weeks apart
  Compare spinal cord fMRI-based response and resting-state functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine T Martucci, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Human Affect & Pain Laboratory (Duke Chronic Pain Lab) — https://anesthesiology.duke.edu/research/martucci-lab
- See also: Please complete this survey as a first step to join the study. — https://redcap.duke.edu/redcap/surveys/?s=RXCMMCPWNKWJELN4